CLINICAL TRIAL: NCT07113275
Title: A National Multicenter, Randomized Controlled Phase III Clinical Trial Comparing Long-Course Versus Short-Course Radiotherapy Followed by Immunotherapy Combined With Total Neoadjuvant Therapy (TNT) to Long-Course Radiotherapy Followed by TNT in High-Risk Locally Advanced Rectal Cancer
Brief Title: A Clinical Trial Comparing Long-Course Versus Short-Course Radiotherapy Followed by Immunotherapy Combined With Total Neoadjuvant Therapy (TNT) to Long-Course Radiotherapy Followed by TNT in High-Risk Locally Advanced Rectal Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, MD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XHZDZLK
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-07

CONDITIONS: Rectal Cancer; Total Neoadjuvant Therapy; Radiotherapy; Immunotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: SCRT + iTNT (Experimental): Group A: SCRT + iTNT
  Radiotherapy (SCRT): Total dose 25 Gy delivered in 5 fractions (5 Gy per fraction, once daily over 5 consecutive days).
  Immunotherapy (HLX10): 300 mg via intravenous infusion every 3 weeks (q3w) for 6 cycles, initiated 1 week after radiotherapy completion.
  Chemotherapy (CAPEOX regimen):
  Oxaliplatin: 130 mg/m² IV infusion over 120 minutes on Day 1.
  Capecitabine: 1000 mg/m² orally twice daily (morning and evening, 30 minutes after meals) on Days 1-14.
  Cycle duration: 3 weeks per cycle; total of 6 cycles during the neoadjuvant phase.
  Then followed by a total mesorectal excision(TME) or Watch & Wait strategy for clinical complete remission voluntary patients.
  Interventions: Radiation: Short-course radiotherapy; Drug: Capecitabine; Drug: Oxaliplatin; Drug: HLX10; Procedure: TME surgery
- Group B: LCRT + iTNT (Experimental): Group B: LCRT + iTNT
  Radiotherapy with Concurrent Chemotherapy (LCRT):
  Total dose 50.4 Gy delivered in 28 fractions (1.8 Gy per fraction, once daily, 5 days per week).
  Concurrent Capecitabine: 825 mg/m² orally twice daily, 5 days per week (administered on radiotherapy days).
  Immunotherapy (HLX10): 300 mg IV infusion q3w for 6 cycles, initiated 2 weeks after radiotherapy completion.
  Chemotherapy (CAPEOX regimen):
  Oxaliplatin: 130 mg/m² IV infusion over 120 minutes on Day 1.
  Capecitabine: 1000 mg/m² orally twice daily (morning and evening, 30 minutes after meals) on Days 1-14.
  Cycle duration: 3 weeks per cycle; initiated 2 weeks post-radiotherapy; total of 6 cycles during the neoadjuvant phase.
  Then followed by a total mesorectal excision(TME) or Watch & Wait strategy for clinical complete remission voluntary patients.
  Interventions: Radiation: Long-course radiotherapy; Drug: Capecitabine; Drug: Oxaliplatin; Drug: HLX10; Procedure: TME surgery
- Group C: LCRT + TNT (Active Comparator): Group C: LCRT + TNT
  Radiotherapy with Concurrent Chemotherapy (LCRT):
  Total dose 50.4 Gy delivered in 28 fractions (1.8 Gy per fraction, once daily, 5 days per week).
  Concurrent Capecitabine: 825 mg/m² orally twice daily, 5 days per week (administered on radiotherapy days).
  TNT Chemotherapy (CAPEOX regimen) with immunotherapy placebo:
  HLX10 placebo: 300 mg IV infusion q3w for 6 cycles, initiated 2 weeks after radiotherapy completion.
  Oxaliplatin: 130 mg/m² IV infusion over 120 minutes on Day 1.
  Capecitabine: 1000 mg/m² orally twice daily (morning and evening, 30 minutes after meals) on Days 1-14.
  Cycle duration: 3 weeks per cycle; initiated 2 weeks post-radiotherapy; total of 6 cycles during the neoadjuvant phase.
  Then followed by a total mesorectal excision(TME) or Watch & Wait strategy for clinical complete remission voluntary patients.
  Interventions: Radiation: Long-course radiotherapy; Drug: Capecitabine; Drug: Oxaliplatin; Procedure: TME surgery; Drug: HLX10 placebo

INTERVENTIONS:
Radiation: Short-course radiotherapy — Eligible subjects will receive short-course radiotherapy (SCRT). One week after the end of treatment, subjects continued to receive neoadjuvant chemotherapy.
  Other Names: SCRT
  Arms: Group A: SCRT + iTNT
Radiation: Long-course radiotherapy — Long-course radiotherapy (LCRT, 50.4 Gy administered in 28 fractions) will be delivered concurrently with oral capecitabine.
  Arms: Group B: LCRT + iTNT; Group C: LCRT + TNT
Drug: Capecitabine — 1000mg/m2, bid, po, d1-14,q3w
Drug: Oxaliplatin — 130mg/m2, ivgtt, d1,q3w
Drug: HLX10 — 300mg, ivgtt, q3w
  Arms: Group A: SCRT + iTNT; Group B: LCRT + iTNT
Procedure: TME surgery — The surgery was performed 1 week after the end of neoadjuvant therapy.
Drug: HLX10 placebo — 300mg, ivgtt, q3w
  Arms: Group C: LCRT + TNT

SUMMARY:
This study is a national multicenter, prospective randomized controlled Phase III clinical trial designed to investigate the potential therapeutic benefit of immunotherapy combined with total neoadjuvant therapy (TNT) and to compare the efficacy of different radiotherapy modalities followed by immunotherapy.

DETAILED DESCRIPTION:
This study is a national multicenter, prospective randomized controlled phase III clinical trial, with the following objectives: 1. For patients with high-risk LARC, to determine whether the efficacy of TNT combined with immunotherapy is superior to that of the treatment mode of LCRT followed by TNT; 2. To compare the differences in efficacy and toxicity between long-course radiotherapy and short-course radiotherapy under the mode of TNT combined with immunotherapy.

For precision management of patients with cCR post-neoadjuvant therapy, dynamic MRD monitoring was implemented, including baseline and follow-up testing for patients having tumors ≤5 cm from the anal verge.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their family members agree to participate in the study and sign the informed consent form;
2. Age 18-75 years, male or female;
3. Histologically confirmed Locally Advanced rectal adenocarcinoma;
4. Immunohistochemistry and/or genetic testing confirmed pMMR/MSS;
5. inferior margin ≤ 10 cm from the anal verge;
6. Pelvic MRI shows high risk [meets one of the following conditions]: • Clinical tumor (cT) staging cT4a or cT4b (according to AJCC 8th Edition) • Extramural vascular infiltration • Clinical lymph node (cN) staging cN2 (according to AJCC 8th Edition) • Mesenteric fascia is involved • Lateral lymph node enlargement
7. ECOG performance status score is 0-1;
8. Untreated with anti-tumor therapy for rectal cancer, including radiotherapy, chemotherapy, surgery, etc;
9. There was no operative contraindication;
10. Laboratory tests were required to meet the following requirements: white blood cell (WBC) ≥ 4×109/L; Absolute neutrophil count (ANC) ≥ 1.5×109/L; Platelet count ≥ 100×109/L; Hemoglobin ≥90 g/L; Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN); Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; Serum creatinine ≤1.5 times the upper limit of normal value or creatinine clearance rate ≥50 mL/min; International normalized ratio (INR) ≤ 1.5 × ULN; Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN;
11. Urinary protein < 2+ or 24-hour urinary protein excretion < 1 g at baseline.

Exclusion Criteria:

1. Patients with non-high-risk pMMR LARC；
2. Subjects who have previously received any form of immunotherapy, including but not limited to immune checkpoint inhibitors, immune checkpoint agonists, immune cell therapy, or any other treatment targeting tumor immunomodulatory mechanisms;
3. Presence of any concurrent disease, condition (including laboratory abnormality), history of substance abuse, or current evidence thereof, which, in the judgment of the Investigator, may compromise subject safety, interfere with the process of obtaining informed consent, affect subject compliance, or confound the safety assessment of the investigational product(s).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Estimated)
Dates: Start 2026-02-11 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) rate | an expected average of 12 months
  Defined as pathological complete response (pCR) + Clinical complete response (cCR)

SECONDARY OUTCOMES:
3-year event-Free Survival | an expected average of 3 years
  The time from the start of treatment to the occurrence of any of the following events, which ever occurs first: tumor disease progression on imaging as assessed by RECIST 1.1; tumor recurrence, including local recurrence or distant recurrence, as assessed on imaging or tissue biopsy transfer; death from any cause.
Overall Survival | an expected average of 5 years
  The time from the date of randomization to the death caused by any cause
Adverse events (AEs) were graded according to the NCI CTCAE version 5·0 | an expected average of 1.5 years
  Adverse events and surgical safety

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Lin, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China